CLINICAL TRIAL: NCT06446167
Title: Comparative Efficacy of Multiwave Locked System Laser, Extracorporeal Shockwave Therapy and Exercise Therapy on Plantar Fasciitis Outcomes: A Randomized Controlled Trial
Brief Title: Comparative Efficacy of Laser, Extracorporeal Shockwave Therapy and Exercise Therapy on Plantar Fasciitis Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Ibrahim Ethem Kirez, Specialist Doctor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: İstanbulSBÜ-FTR-IEK-01
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Plantar Fascitis
Keywords: Plantar Fasciitis; Exercise; Lasers; Extracorporeal Shockwave Therapy
MeSH Terms: conditions — Fasciitis, Plantar; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 60 patients met the eligibility criteria and were enrolled in the study. The eligible participants were randomized into three distinct groups each comprising 20 individuals: an exercise alone group (Exercise group), an exercise combined with MLS laser therapy group (Laser group), and an exercise combined with ESWT group (ESWT group). Randomization was conducted using a computer-assisted program
Who Masked: Outcomes Assessor
Masking Description: The evaluation of outcomes was performed by an assessor blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise group (Active Comparator): All groups received a regimen of daily exercises, including stretches for the plantar fascia and Achilles tendon, and strengthening exercises for the calf muscles and foot intrinsic muscles. Each type of exercise was demonstrated to the participants by the same physiotherapist at the beginning of the treatment process, to be performed twice a day with 10 repetitions each time.
  Interventions: Other: Exercises
- Laser group (Active Comparator): The MLS Laser applied to the treatment group was administered using an ASA brand Mphi model device. Patients in the Laser group were positioned in a prone position. Treatment was applied continuously for 7 minutes along the plantar fascia, sole of the foot, heel area, and Achilles tendon in accordance with the plantar fasciitis treatment program on the device, at a dose of 1.73 J/cm2 and a frequency of 700 Hz. A treatment program was established with 3 sessions per week, totaling 10 sessions. Patients receiving laser therapy also continued with their exercise programs.
  Interventions: Other: Exercises; Other: MLS Laser Treatment
- ESWT group (Active Comparator): The treatment group was administered with the Swiss DolorClast Master ESWT device, which produces radial shock waves. Patients in the ESWT group were positioned in a prone position. The most painful point in the heel area was identified through palpation. Gel was applied to this area, followed by the surrounding soft tissues, towards the plantar fascia and the attachment area of the Achilles tendon at the dorsal aspect of the heel. Radial ESWT treatment was applied at a frequency of 10 Hz, pressure of 2.5 bars, and 2000 impulses per session, once a week for a total of 4 sessions. Patients receiving ESWT therapy also continued with their exercise programs.
  Interventions: Other: Exercises; Other: ESWT treatment

INTERVENTIONS:
Other: Exercises — All groups received a regimen of daily exercises, including stretches for the plantar fascia and Achilles tendon, and strengthening exercises for the calf muscles and foot intrinsic muscles. Each type of exercise was demonstrated to the participants by the same physiotherapist at the beginning of the treatment process, to be performed twice a day with 10 repetitions each time.
Other: MLS Laser Treatment — The MLS Laser applied to the treatment group was administered using an ASA brand Mphi model device. Patients in the Laser group were positioned in a prone position. Treatment was applied continuously for 7 minutes along the plantar fascia, sole of the foot, heel area, and Achilles tendon in accordance with the plantar fasciitis treatment program on the device, at a dose of 1.73 J/cm2 and a frequency of 700 Hz. A treatment program was established with 3 sessions per week, totaling 10 sessions
  Arms: Laser group
Other: ESWT treatment — The treatment group was administered with the Swiss DolorClast Master ESWT device, which produces radial shock waves. Patients in the ESWT group were positioned in a prone position. The most painful point in the heel area was identified through palpation. Gel was applied to this area, followed by the surrounding soft tissues, towards the plantar fascia and the attachment area of the Achilles tendon at the dorsal aspect of the heel. Radial ESWT treatment was applied at a frequency of 10 Hz, pressure of 2.5 bars, and 2000 impulses per session, once a week for a total of 4 sessions
  Arms: ESWT group

SUMMARY:
This study aims to evaluate the effectiveness of exercise combined with ESWT (Extracorporeal Shockwave Therapy), exercise combined with MLS (Multiwave Locked System) laser therapy, and exercise alone in female patients diagnosed with unilateral plantar fasciitis, using Visual Analog Scale (VAS), Heel Tenderness Index (HTI), Foot and Ankle Outcome Score (FAOS), Foot Function Index (FFI) and fall risk, as clinical parameters to assess any differences in effectiveness levels among these treatments.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a prevalent condition characterized by the degeneration of the plantar fascia, a band of connective tissue that originates from the calcaneus to the proximal phalanges and the skin of the foot's anterior part. Despite common misconceptions, plantar fasciitis is not primarily an inflammatory process but results from repetitive microtears leading to a secondary inflammatory reaction of the plantar fascia.

Despite the condition's self-limiting nature, with 70% to 80% of patients experiencing symptom relief through conservative treatment alone, a combination of treatments is often necessary for many. Conservative interventions include rest, cold application, stretching and strengthening exercises, orthotic devices, lifestyle modifications, weight loss, and night splints. Additionally, non-invasive physical therapy modalities such as Extracorporeal Shock Wave Therapy (ESWT), laser, and ultrasound have shown to be cost-effective and accessible treatment options. Invasive treatments, including injections and surgery, are considered for resistant cases

Previous studies have examined the effectiveness of ESWT, Low level laser therapy, High intensity laser therapy, and exercise treatments in patients with PF, demonstrating their efficacy. Although there are studies investigating the effectiveness of MLS laser therapy on various musculoskeletal pathologies, to our knowledge, there is no study specifically examining its efficacy on PF

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Female gender
* Symptoms persisting for at least 6 weeks
* Unilateral plantar fasciitis
* Consent to participate in the study

Exclusion Criteria:

* Male gender
* Bilateral plantar fasciitis
* Treatment with ESWT, laser or injection therapy for plantar fasciitis in the previous year
* Participation in a physical therapy program for plantar fasciitis in the last six months
* History of systemic inflammatory disease
* History of lower extremity fracture or surgery
* Pregnancy
* History of epilepsy
* Malignancy
* Active infection
* Coagulation disorders
* Severe cardiac disease or history of pacemaker
* History of neuromuscular disease affecting balance parameters
* Regular use of nonsteroidal antiinflammatory drugs

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | one month
  VAS is a scale 10 cm in length, starting from "no pain" and ending with "unbearable pain" (0: no pain, 10: unbearable pain). Patients indicate the severity of their pain by marking the appropriate point on this scale. The distance between "no pain" and this marked point is measured and recorded in centimeters

SECONDARY OUTCOMES:
Foot Function Index (FFI) | one month
  The FFI is a self-reported questionnaire designed to assess the impact of foot pathology on three domains: pain (9 items), disability (9 items), and activity limitation (5 items). Each item is rated on a scale from 0 (no issue) to 10 (severe issue). The scores are normalized to a 100-point scale for each domain, offering a detailed metric for functional impairment. To calculate the Total FFI score, the average of the scores from the three subheadings is taken. Higher scores are associated with more severe illness. The Turkish adaptation of the FFI was conducted by Yalıman et al.
Foot and Ankle Outcome Score (FAOS) | one month
  Adapted from the knee injury and osteoarthritis outcome score, the FAOS is a detailed tool that evaluates five domains: symptoms and stiffness (7 items), pain (9 items), daily living activities (17 items), sports and recreational activities (5 items), and quality of life (4 items). Each question has 5 different responses that can be scored from 0 for the best condition to 4 for the worst condition, based on the intensity of the complaint. The result ranges from 0 to 100. A score of 0 indicates the worst possible foot and ankle symptoms, while a score of 100 indicates no foot and ankle symptoms. The Total FAOS score is calculated by taking the percentage of responses given to all 42 questions, regardless of the subheadings. The Turkish adaptation of the FAOS was conducted by Karatepe et al. in 2009.
Heel Tenderness Index (HTI) | one month
  The HTI quantifies pain sensitivity in the heel through clinical palpation. It is scored from 0 (no pain) to 3 (severe pain with withdrawal reflex), enabling objective assessment of localized tenderness.
Biodex Fall Risk Assessment | one month
  The Biodex balance system SD-2014 is a robotic device equipped with computer software that allows tilting up to 20° in all directions, enabling objective assessment of balance and fall risk. High scores indicate impaired balance and increased risk of falling. During measurement, patients are asked to remove their shoes and step onto the platform, maintaining a comfortable position while visually monitoring themselves on the screen to stay centered. Patients are instructed to maintain this position throughout the measurements. Subsequently, according to the fall risk measurement protocol of the device, fall risk calculations are performed at levels 12-8, with 20-second test durations repeated 3 times. The fall risk resulting from these 3 measurements is provided as the overall stability index (OSI) score.

CONTACTS AND LOCATIONS:
Overall Officials: İbrahim Ethem Kirez, Principal Investigator — İstanbulSBÜ
Locations (1):
- İstanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No